CLINICAL TRIAL: NCT03059368
Title: New Bone Fixation Plate for the Repair of Tibial Avulsion Fracture of Posterior Cruciate Ligament of the Knee: a Prospective, Open-label, Self-controlled, Clinical Trial
Brief Title: New Bone Fixation Plate for the Repair of Tibial Avulsion Fracture of Posterior Cruciate Ligament of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cangzhou Central Hospital (Other)
Responsible Party: Principal Investigator, Guangdong Chen, Attending Physician, Cangzhou Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CangzhouCH_01
Record Dates: First submitted 2017-02-12; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Tibial Fractures
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- new bone fixation plate with screw (Experimental): Fracture ends and injured posterior cruciate ligament will be exposed in twenty patients with tibial avulsion fracture of posterior cruciate ligament of knee through posterior approach. Open reduction will be conducted. The posterior cruciate ligament will be reconstructed with a new bone fixation plate with screw(cancellous bone screw).
  Interventions: Device: new bone fixation plate with screw

INTERVENTIONS:
Device: new bone fixation plate with screw — Fracture ends and injured posterior cruciate ligament will be exposed in twenty patients with tibial avulsion fracture of posterior cruciate ligament of knee through posterior approach. Open reduction will be conducted. The posterior cruciate ligament will be reconstructed with a new bone fixation plate with screw(cancellous bone screw).

SUMMARY:
To construct a self-designed plate fixation device for posterior cruciate ligament reconstruction, aim to verify its advantages on anatomical knee stability, so as to achieve fracture healing and keep tension after posterior cruciate ligament reconstruction.

DETAILED DESCRIPTION:
History and current related studies Posterior cruciate ligament of the knee is an important structure to maintain stability of the knee, and can prevent backward displacement of the tibia, so the violence that causes the tibia to move backward can cause posterior cruciate ligament rupture. Tibial avulsion fracture of posterior cruciate ligament of the knee will lead to unstable posterior movement and rotation of the knee and accelerate the degeneration of the knee. Thus, maintaining the tension of posterior cruciate ligament and restoring anatomical stability of the knee affect early rehabilitation and surgical treatment, and are the difficulty and key point of sports medicine.

When tibial avulsion fracture of posterior cruciate ligament of knee is treated with open reduction and rivet fixation, hollow screw fixation or arthroscopic reconstruction of the posterior cruciate ligament, plaster fixation is often required for flexion and extension exercises. However, the importance of early tension reconstruction of posterior cruciate ligament is often ignored. How to select the fixation method for tibial avulsion fracture of posterior cruciate ligament and how to restore the anatomical stability of the joint are still controversial. In recent years, with the development of surgical techniques and instruments and the popularization of the concept of precision surgical treatment, high requirements are put forward for the new fracture fixation methods.

Data collection, management, analysis, open access

1. Data collection: Case report forms will be collected, processed using Epidata software (Epidata Association, Odense, Denmark), collated, and then recorded electronically by data managers using a double-data entry strategy.
2. Data management: The locked electronic database will be accessible and locked only by the project manager. This arrangement will not be altered. The Cangzhou Central Hospital, China will preserve all of the data regarding this trial.
3. Data analysis: A professional statistician will statistically analyze the electronic database and will create an outcome analysis report that will be submitted to the lead researchers. An independent data monitoring committee will supervise and manage the trial data, ensuring a scientific and stringent trial that yields accurate and complete data.
4. Data open access: Anonymized trial data will be published at www.figshare.com.

Statistical analysis

1. Statistical analysis will be performed using SPSS 13.0 software (SPSS, Chicago, IL, USA) and will follow the intention-to-treat principle. Normally distributed measurement data will be expressed as means ± standard deviation and minimums and maximums. Non-normally distributed measurement data will be expressed as the lower quartile (q1) and median and upper quartiles (q3). The count data will be expressed as a percentage.
2. Normally distributed data of HSS and Lysholm Knee Scoring Scale scores at preoperative, postoperative 3 and 12 months will be analyzed with one-way analysis of variance and least significant difference. Non-normally distributed data will be analyzed using Kruskall-Wills H test and Cohen's d test. Patient satisfaction and incidence of adverse reactions at postoperative 3 and 12 months will be compared using McNemar χ2 test. The significance level will be α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Tibial avulsion fracture of posterior cruciate ligament of knee
* Limitation of flexion and extension of knee, posterior drawer test (+)
* History of knee trauma
* An age of 35-58 years
* Irrespective of gender
* Signed informed consent

Exclusion Criteria:

* Pathologic fracture
* Fracture accompanied by nerve injury
* Knee osteoarthritis
* Other chronic knee diseases

Ages: 35 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Hospital for Special Surgery Knee Score | changes of baseline, postoperative month 3 and month 12
  To evaluate knee function. The higher the score, the better the recovery of knee function is.

SECONDARY OUTCOMES:
Lysholm Knee Scoring Scale | changes of baseline, postoperative month 3 and month 12
  To evaluate knee function. The higher the score, the better the recovery of knee function is.
Patient satisfaction | changes of postoperative month 3 and month 12
  The percentage of the number of patients with satisfactory knee function to the total number of cases. The higher the value, the more satisfied with the treatment plan.

CONTACTS AND LOCATIONS:
Overall Officials: Guangdong Chen, Master, Principal Investigator — Cangzhou Central Hospital

IPD SHARING:
Plan to Share IPD: Undecided